CLINICAL TRIAL: NCT05804526
Title: An Open-label, Non-randomised, Multi-center Study to Evaluate the Safety， and Efficacy Off RC88 Combined With Sintilimab in AdvancedSolid Tumours
Brief Title: A Study of RC88 Combined With Sintilimab for Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC88 C003
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumours
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC88+Sintilimab Injection (Experimental): RC88+Sintilimab Injection Arm
  Interventions: Drug: RC88; Drug: Sintilimab Injection

INTERVENTIONS:
Drug: RC88 — 1.5mg/kg ，2.0mg/kg ，2.5mg/kg by intravenous (IV) infusion，every 3 weeks
Drug: Sintilimab Injection — Sintilimab 200mg by intravenous (IV) infusion，every 3 weeks
  Other Names: Sintilimab

SUMMARY:
This study will evaluate safety , clinical pharmacology and efficacy of intravenous RC88 combined with Sintilimab in advancedsolid tumours

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consen
2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
3. Predicted survival ≥ 12 weeks
4. Phase I (Phase I) was included and confirmed as MSLN positive (≥1+ after IHC test by central laboratory).Failure, intolerance, or lack of standard treatment has been identified by tissue or cytology The MSLN test is not required for patients with advanced malignant tumor and for subjects diagnosed with malignant mesothelioma;
5. Adequate organ function required
6. Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.

Exclusion Criteria:

1. Cancer metastases in the brain
2. Active infection or past hepatitis B or C infection
3. Major surgery less than 1 month before the start of the study
4. Uncontrolled heart disease
5. History of allergy to mesothelin-directed antibodies, tubulysin, monoclonal antibodies related compounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
RP2D | 28 days after first treatment
  Incidence of DLT (dose limiting toxicity) of RC88 combined with Sintilimab

SECONDARY OUTCOMES:
ORR | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Maximum Concentration (Cmax) of RC88 | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 24, 48, 96, 168 hours
  Dose Escalation and Expansion Part
Progression Free Survival (PFS) | 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuankai, M.D., Study Director — Leading PI
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No